CLINICAL TRIAL: NCT06111300
Title: The Effect of Dexmedetomidine on the Incidence of Post-operative Delirium in Elderly Patients Undergoing Emergency Laparotomy
Brief Title: Dexmedetomidine Effect on Delirium of Elderly Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Ahmed Gharib Ahmed, assisstant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: delirium in elderly patients
Record Dates: First submitted 2023-10-11; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Delirium in Old Age
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Group D (dexmedetomidine group): Patients in this group will receive loading dose of dexmedetomidine 0.7 ug/kg over 10 min. then maintenance dose 0.2 - 1 ug/kg/hr till end of surgery.Group C (control group): Patients in this group will receive volum- matched normal saline infusion (NaCL 0.9%) as a placebo.
Who Masked: Participant
Masking Description: control group will take placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group d (Experimental): Patients in this group will receive loading dose of dexmedetomidine 0.7 ug/kg over 10 min. then maintenance dose 0.2 - 1 ug/kg/hr till end of surgery.
  Interventions: Drug: Dexmedetomidine
- group c (Placebo Comparator): Patients in this group will receive volume- matched normal saline infusion (NaCL 0.9%) as a placebo.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Group D (dexmedetomidine group): Patients in this group will receive loading dose of dexmedetomidine 0.7 ug/kg over 10 min. then maintenance dose 0.2 - 1 ug/kg/hr till end of surgery. Group C (control group): Patients in this group will receive volum- matched normal saline infusion (NaCL 0.9%) as a placebo.

SUMMARY:
The Effect of Dexmedetomidine on the Incidence of Delirium Incidence of Post-operative Delirium in Elderly Patients Undergoing Emergency Laparotomy

DETAILED DESCRIPTION:
Delirium is an acute brain illness, which involves changes in consciousness, attention, cognition, and perception. Delirium is a common postoperative complication, especially in older patients, and is an independent predictor for postoperative mortality. It may put patients at risk of post-operative cognitive dysfunction (POCD) , Conversion rates to dementia up to 70% have been demonstrated in patients who are aged ≥ 65 y.The incidence of postoperative delirium ranges from 5% to 51% For major open abdominal surgery. Post-operative delirium (POD) is associated with: increased mortality; prolonged hospital stay; and major peri-operative complications and morbidity. For every day of postoperative delirium on the ICU, 1-year survival probability decreases by approximately 10%. it has multiple associated features including altered arousal, disorganised thinking, perceptual disturbances, psychosis, and sleep-wake cycle disturbance. Delirium occurs in patients of all ages but the highest incidence is in older people with a background of chronic central nervous system (CNS) disease. Several hypotheses describe different aspects of the pathophysiology of delirium; Increased Age: lead to diminished physiologic reserve and increased vulnerability to physical stress, decreased brain blood perfusion, increased neuron loss, and changes in the proportion of stress-regulating neurotransmitters. Neuroinflammation: Peripheral inflammatory insults damage endothelial cell-cell adhesions at the blood-brain barrier. The increased endothelial permeability promotes inflammation in the central nervous system, causing further damage, ischemia, and neuronal death.Reactive Oxidation Species: are a mediator of cellular damage due to its high lipid content and low antioxidant capacity.Circadian Rhythm Dysregulation: Disruption in sleep duration leads to dysfunction of many systems including regulation of sleep-wake cycles, glucose regulation, core body temperature, antioxidant defenses, and immune system response.Neurotransmitter Imbalance: Delirium is associated with decreased acetylcholine and increased dopamine activity. Neuroendocrine: Increased glucocorticoid release in response to physiologic stress increases the vulnerability of neurons to subsequent damage and impacts the regulation of gene transcription, cellular signaling, and glial cell behavior.Management of deliriumNon-pharmacologic interventions; which are the main treatments for delirium : Decreasing environmental disturbances, increase uninterrupted sleep by use of eyeglasses or hearing aids to optimize hearing and vision, use of tools to improve orientation including clocks and calendars, frequent mobilization.pharmacologic therapies such as; Benzodiazepines, Antipsychotics and Other medications include; haloperidol, quetiapine, and risperidone.Dexmedetomidine is a highly potent a2-agonist, which is used widely in critical care for delirium symptom control. It is known for its sparing properties on delirogenic medication such as sedatives and opioids. Furthermore, it displays antisympathetic, co-analgesic, anxiolytic and sedative effects with minimal respiratory depression. These effects are likely mediated by centraly inhibitive effects of dexmedetomidine on the nucleus coeruleus in the brain.Recent meta-analyses show a significantly lower incidence of delirium for dexmedetomidine when given intra- and postoperatively. Peng et al. also found a significant reduction in 30-day mortality and ICU and hospital stay in cardiac surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 60 years or older of either gender.

  * Patient undergoing emergency laparotomy either trauma or non-trauma patients.

Exclusion Criteria:

* • Patients unable to provide written consent.

  * Patients less than 60 years.
  * Known drug intolerance or allergy to dexmedetomidine.
  * Patients previously diagnosed to suffer from major neurocognitive disorder, defined by a mini-mental state examination (MMSE) score < 24.
  * Severe audiovisual impairment.
  * Child C chronic liver disease.
  * Traumatic brain injury.
  * Intracranial bleeding < 1y.
  * Psychiatric illness.
  * History of alcohol or drug abuse.
  * Preoperative cerebrovascular accident with residual neurological deficit.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Delirium among elderly | 3 days
  Incidence of delirium among elderly patients undergoing emergency laparotomy.

IPD SHARING:
Plan to Share IPD: No